CLINICAL TRIAL: NCT06380725
Title: A Randomized, Double-blind Placebo Controlled Trial of High Intensity Transcranial Current Stimulation in Patients With Alzheimer's Disease
Brief Title: The Treatment of High Intensity Transcranial Current Stimulation for Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Jiong Shi, Director, Principal Investigator, Clinical Professor, Anhui Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: jshim8zay6vd
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Dementia
Keywords: Alzheimer's Disease; biomarker; Transcranial alternating current stimulation; functional connectivity; Brain network
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: Investigators designed a randomized double-blinded placebo-controlled trial by randomly dividing subjects into two groups: one is the treatment group and the other is the placebo group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigators designed a double-blinded trial in which neither the investigator nor the subjects know whether they will be received the treatment or a placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- control group (Placebo Comparator): Subjects sit comfortably in a recliner and receive FDA-approved transcranial alternating current stimulation (sham stimulation) with trained operators following standardized instructions. Subjects are advised to relax, drink water, and even sleep, and not communicate with the operator as much as possible.
  Interventions: Device: Transcranial alternating current stimulation(sham stimulation)
- treatment group (Experimental): Subjects sit comfortably in a recliner and receive FDA-approved transcranial alternating current stimulation (real stimulation) with trained operators following standardized instructions. Subjects are advised to relax, drink water, and even sleep, and not communicate with the operator as much as possible.
  Interventions: Device: Transcranial alternating current stimulation(real stimulation)

INTERVENTIONS:
Device: Transcranial alternating current stimulation(real stimulation) — Real tACS is an emerging noninvasive neuro-regulation technique that applies a specific frequency of stimulation and a specific intensity of weak current to the brain by means of electrodes placed in the skull.
  Arms: treatment group
Device: Transcranial alternating current stimulation(sham stimulation) — Transcranial alternating current stimulation (sham-stimulation) is an emerging noninvasive neuro-regulation technique that applies a specific frequency of stimulation and a specific intensity of a weak current to the brain by means of electrodes placed in the skull. The subjects felt the same as the real stimulus when receiving the sham-stimulus treatment, but the sham-stimulus did not have the current stimulation.
  Arms: control group

SUMMARY:
Alzheimer's disease (AD) is a neurodegenerative disorder characterized by progressive cognitive dysfunction and behavioral impairment. It is currently the most common type of dementia in the old age. At present, the clinical treatment of Alzheimer's disease is expensive and has side effects, so it is very important to explore new methods of treatment for AD. Investigators designed a prospective, randomized, double-blinded and placebo-controlled trial to investigate the effect of transcranial alternating current stimulation (tACS) on cognitive function in AD patients and to assess the biological effectiveness of the treatment.

DETAILED DESCRIPTION:
As the population is aging, there is an urgent need to develop new methods of treatment for AD. Noninvasive neuro-regulation is a new technique in treating neuropsychiatric diseases. It include transcranial magnetic stimulation, traditional transcranial direct current stimulation, traditional transcranial alternating current stimulation and etc. Previously, conventional transcranial direct current stimulation had shown inconsistent results in the treatment for AD. This may be related to the low current density of traditional electrical stimulation in deep brain areas, such as hippocampus and amygdala, and leading to poor stimulation effect. Compared with the traditional transcranial electrical stimulation technology, the high intensity tACS greatly improves the current intensity, so that the electric field intensity to the deep brain nucleus during stimulation is greatly increased, and it avoids side effects such as burning sensation. Therefore, it could be used for AD patients. However, there are few clinical studies on high intensity tACS on AD, so investigators designed a randomized double-blinded placebo-controlled trial to explore the effect of high-current tACS on AD. At the same time, multimodal functional brain imaging before and after treatment will be used to compare the changes of brain function activation and cerebral hemodynamics in AD.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of National Institute on Aging and Alzheimer's Association (NIA-AA) 2011 for Alzheimer's disease, Clinical Dementia Rating (CDR) score is greater than or equal to 0.5 and less than or equal to 1, and amyloid PET imaging is positive.
2. Have the ability to cooperate with neuropsychological testing, EEG measurement, and MRI examination;
3. Have willingness to undergo cognitive psychological evaluation;
4. Do not have cognitive impairment due to other degenerative diseases or viral and immune encephalitis;
5. The length of schooling is at least 3 years.

Exclusion Criteria:

1. Do not suffer from severe depression, anxiety and other mental illness;
2. Do not suffer from major diseases such as tumors, heart and lung diseases, nervous system diseases, etc.
3. Do not have been diagnosed with other dementia such as Parkinson's disease dementia (PDD), frontotemporal dementia (FTD), lewy body dementia (DLB), and normal cranial pressure hydrocephalus (NPH).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive appraisal | A total of 5 times will be measured, before the treatment, immediately after the treatment, 1-, 3- and 6-month follow-ups.
  A series of cognitive functions such as verbal function and visuospatial functions will be evaluated by Clock drawing test (maximum score =4, minimum score =0, the higher the better) and Boston Naming Test (maximum score =30, minimum score =0, the higher the better) ect.
Global Cognitive appraisal | A total of 5 times will be measured, before the treatment, immediately after the treatment, 1-, 3- and 6-month follow-ups.
  Overall cognitive function will be assessed through Clinical Dementia Rating(maximum score =3, minimum score =0, the higher the better) and Minimum Mental State Examination(maximum score =30, minimum score =0, the higher the better) ect.
Psychobehavioral assessment | A total of 5 times will be measured, before the treatment, immediately after the treatment, 1-, 3- and 6-month follow-ups.
  The mental and behavioral states of the patients will be evaluated by Neuropsychiatric Inventory(maximum score =144, minimum score =0, the lower the better) and Hamilton's Depression Scale (maximum score =68, minimum score =0, the lower the better) ect.

SECONDARY OUTCOMES:
Near-infrared spectroscopy | A total of 5 times will be measured, before the treatment, immediately after the treatment, 1-, 3- and 6-month follow-ups.
  The brain function of the patients before and after treatment will be assessed by near infrared functional brain imaging
Event related potential measurement | A total of 5 times will be measured, before the treatment, immediately after the treatment, 1-, 3- and 6-month follow-ups.
  Event related potential indicators will be evaluated before and after treatment by electroencephalogram.
Peripheral blood biomarkers | A total of 5 times will be measured, before the treatment, immediately after the treatment, 1-, 3- and 6-month follow-ups.
  Peripheral blood biomarkers such as the concentration of tau and amyloid protein will be detected by SiMoA before and after treatment
Magnetic Resonance Imaging | A total of 3 measurements, before treatment, immediately after treatment, 1 month follow-up
  Brain function before and after treatment will be measured by MRI
Incidence of side effects | Interviews will be conducted daily after treatment and once at 1-, 3- and 6-month follow-ups.
  After daily treatment, the subjects will be interviewed by the investigator, and the possible adverse reactions such as headache and fatigue ect. observed will be collected and recorded in the case report form. After the end of the experiment, investigators will calculate the probability of the occurrence of the side effects observed in the experiment through the case report form in the interview.

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Shi, doctor, Study Chair — The First Affiliated Hospital of University of Science and Technology of China

IPD SHARING:
Plan to Share IPD: Yes
After the research is published in an academic journal, a link to the laboratory website will be provided in the article so that others can view supplementary materials, etc. Access to the data requires the consent of the principal investigator and the ethics committee.
Supporting Information: Study Protocol
Time Frame: After the research is published in an academic journal, a link to the laboratory website will be provided in the article.
Access Criteria: Access to the data requires the consent of the principal investigator and the ethics committee.